CLINICAL TRIAL: NCT06286098
Title: Effect of Alpha Lipoic Acid on the Clinical Outcome of Pediatric Patients Undergoing Hemodialysis
Brief Title: Alpha Lipoic Acid in Pediatrics on Hemodialysis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Eva Pharma (Industry)
Responsible Party: Principal Investigator, mahmoud mohsen, Researcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ALA in Pediatrics on HD
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis Complication; Pediatric Kidney Disease; Cardiovascular Complication
Keywords: Alpha Lipoic Acid; alpha-lipoic acid; Thioctic acid; Hemodialysis; E-selectin; eselectin; Children Kidney
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Alpha lipoic acid) Active Group (Experimental): Alpha Lipoic Acid orally along with the standard care of therapy for a duration of 6 months.
  Dose: 600 mg once daily.
  Interventions: Drug: Alpha lipoic acid
- (Placebo) Control Group (Placebo Comparator): Placebo along with the standard care of therapy for a duration of 6 months.
  Dose: One Tablet daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alpha lipoic acid — THIOTACID 600 MG ORIGINAL ® Tablets manufactured by EVA PHARMA
  Other Names: Thioctic Acid
  Arms: (Alpha lipoic acid) Active Group
Other: Placebo — Placebo identical Tablets are manufactured by EVA PHARMA containing the same excipients without Alpha Lipoic Acid.
  Arms: (Placebo) Control Group

SUMMARY:
The goal of this clinical trial is to test alpha lipoic acid in children undergoing hemodialysis. The main questions it aims to answer are:

* Will the use of alpha lipoic acid lower cardiovascular events in that population?
* Is the incidence of those cardiovascular events linked to the oxidative stress and endothelial dysfunction in that population?
* Will the drug cause side effects?

Participants will:

* take either one dose daily of 600mg tablet Alpha lipoic acid orally or a look-alike tablet containing no drug.
* be monitored for the occurrence of cardiovascular events (stroke, angina, etc.)
* be monitored for the occurrence of side effects
* give blood samples for testing serum levels of E-selectin biomarker and superoxide dismutase enzyme
* undergo clinical examinations (Echocardiogram, Duplex ultrasonography, Intima-Media-Thickness) Researchers will compare between the group taking alpha lipoic acid and the group taking the look-alike tablet.

DETAILED DESCRIPTION:
A Double-Blinded, Paralleled, Randomized, Placebo-Controlled Clinical Trial will be conducted at the Pediatric Nephrology and Dialysis Unit, Children's Hospital, Ain Shams University, Cairo, Egypt to detect the efficacy of alpha lipoic acid in reducing cardiovascular events by reducing oxidative stress-mediated endothelial dysfunction in pediatric population on regular hemodialysis by assessment of:

1. E-selectin as an Endothelial biomarker
2. SOD as an Oxidative stress biomarker
3. Indicators of CVS dysfunction by;

   * Duplex ultrasonography
   * Echocardiogram with stress on Ejection Fraction
   * Intimal medial thickness
4. Occurrence of CVS events

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants admitted to Pediatric Hemodialysis Unit for regular hemodialysis.
* The ability to swallow capsules will be enrolled in the study.

Exclusion Criteria:

* Participants who suffered from severe congestive heart failure
* Participants suffering from inflammatory diseases or other diseases that may increase oxidative stress.
* Participants taking supplements that decrease oxidative stress or inflammatory markers
* Participants with hypersensitivity to alpha lipoic acid
* Participants who are non-compliant.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Serum level of E-Selectin | at baseline and after the duration of treatment (6 months)
  The effect of ALA supplementation on the serum level of E-Selectin in pediatric patients on regular hemodialysis.

SECONDARY OUTCOMES:
Serum levels of superoxide dismutase (SOD) | at baseline and after the duration of treatment (6 months)
  The effect of ALA supplementation on the serum level of SOD in pediatric patients on regular hemodialysis.
Number of cardiovascular events | for the duration of treatment (6 months)
  Counting the number of cardiovascular events (stroke, angina, etc.) through monitoring
Number of Adverse effects | for the duration of treatment (6 months)
  Evaluation of the safety of ALA supplementation in pediatric hemodialysis patients in terms of proportion of adverse drug events and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Mohsen, Pharmacist, Principal Investigator — Misr University for Science and Technology
Locations (1):
- New Pediatrics Hospital, Faculty of Medicine, Ain Shams University, Cairo, El Weili, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fogacci F, Rizzo M, Krogager C, Kennedy C, Georges CMG, Knezevic T, Liberopoulos E, Vallee A, Perez-Martinez P, Wenstedt EFE, Satrauskiene A, Vrablik M, Cicero AFG. Safety Evaluation of alpha-Lipoic Acid Supplementation: A Systematic Review and Meta-Analysis of Randomized Placebo-Controlled Clinical Studies. Antioxidants (Basel). 2020 Oct 19;9(10):1011. doi: 10.3390/antiox9101011. PMID 33086555
- [Background] Haghighatdoost F, Hariri M. The effect of alpha-lipoic acid on inflammatory mediators: a systematic review and meta-analysis on randomized clinical trials. Eur J Pharmacol. 2019 Apr 15;849:115-123. doi: 10.1016/j.ejphar.2019.01.065. Epub 2019 Feb 2. PMID 30721699
- [Background] Huang EA, Gitelman SE. The effect of oral alpha-lipoic acid on oxidative stress in adolescents with type 1 diabetes mellitus. Pediatr Diabetes. 2008 Jun;9(3 Pt 2):69-73. doi: 10.1111/j.1399-5448.2007.00342.x. Epub 2008 Jan 22. PMID 18221433
- [Background] Li LC, Tain YL, Kuo HC, Hsu CN. Cardiovascular diseases morbidity and mortality among children, adolescents and young adults with dialysis therapy. Front Public Health. 2023 Apr 12;11:1142414. doi: 10.3389/fpubh.2023.1142414. eCollection 2023. PMID 37124791
- [Background] Malatino LS, Stancanelli B, Cataliotti A, Bellanuova I, Fatuzzo P, Rapisarda F, Leonardis D, Tripepi G, Mallamaci F, Zoccali C. Circulating E-selectin as a risk marker in patients with end-stage renal disease. J Intern Med. 2007 Oct;262(4):479-87. doi: 10.1111/j.1365-2796.2007.01841.x. PMID 17875185
- [Background] Al-Nami MS, Al-Kuraishy HM, Al-Gareeb AI. Impact of thioctic acid on glycemic indices and associated inflammatory-induced endothelial dysfunction in patients with type 2 diabetes mellitus: A case control study. Int J Crit Illn Inj Sci. 2020 Sep;10(Suppl 1):21-27. doi: 10.4103/IJCIIS.IJCIIS_62_19. Epub 2020 Sep 16. PMID 33376686